CLINICAL TRIAL: NCT04117815
Title: Hair-Safe Study: Scalp Cooling for Hair Saving in Women Undergoing Chemotherapy
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: 1049/2018
Record Dates: First submitted 2019-06-17; First posted 2019-10-07 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer Female; Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- study group: Patients with breast or gynecological cancer planning to undergo chemotherapy Chemotherapy can be neoadjuvant, adjuvant or palliative Up to two lines of chemotherapy are allowed. Adjuvant therapy counts as one line.
  Chemotherapy regime is associated with alopecia. Chemotherapy must be planned for at least 4 cycles of taxane or antracycline- based chemotherapy regimen No alopecia of any reason (up-front) No overt cognitive impairment and fluent in German Written informed consent Age 18 and older
  Interventions: Device: Paxman Scalp Cooling System; Other: Alopecia Assessments
- reference group: For the purpose of comparison, a reference sample will be included in the study applying to the following inclusion criteria:
  Patients with breast or gynecological cancer planning to undergo chemotherapy Chemotherapy can be neoadjuvant, adjuvant or palliative Up to two lines of chemotherapy are allowed. Adjuvant therapy counts as one line.
  Chemotherapy regime is associated with alopecia. Chemotherapy must be planned for at least 4 cycles of taxane or antracycline- based chemotherapy regimen Refuse to undergo scalp cooling Patients who have been excluded for the study group for the reason of migraine Written informed consent Age 18 and older
  Patients from the reference group complete the same survey as the study group. Group comparisons will be adjusted for baseline body image and reasons for refusal.
  Interventions: Other: Alopecia Assessments

INTERVENTIONS:
Device: Paxman Scalp Cooling System — All patients who accomplish inclusion criteria and do not exhibit any contraindication undergo scalp cooling with the following conditions:
  * Minimum 30 minutes pre-infusion cooling
  * Cooling for the duration of chemotherapy infusion
  * Minimum 90 minutes post-infusion cooling Scalp cooling is performed within the study group at each CT session.
  Groups: study group
Other: Alopecia Assessments — Patients (study group and reference group) will be assessed at the following time Points:
  * Baseline
  * at the half-way Point of the cyles
  * at the last CT cycle
  * 3 months after completion of Treatment
  * 6-9 months after treatment completion
  The assesments include the following
  * Photographs of the head, which are evaluated using the CTCAEv4.0
  * Questionnaire including the NCI- PRO-CTCAE-ITEMS, EORTC QLQ-C30, EORTC QLQ-B23, Body Image Scale, PRO-CTACAEs and Hairdex questionnaire

SUMMARY:
Chemotherapy (CT) is a frequent and well established treatment in women with breast and gynecological tumors. Alopecia is one of the most common side effects of CT seriously impairing patient quality of life and body image. While other CT associated side effects can be controlled by supportive treatment strategy, adequate preventive measures for alopecia have been lacking. New evidence supports the efficacy of scalp cooling for alopecia prevention during CT.

DETAILED DESCRIPTION:
Scalp cooling using cooling caps has been identified as an effective treatment option against CT-induced alopecia in numerous European countries. Originally, crashed ice was used to cause vasoconstriction and consequently diminish CT uptake to hair follicles during CT. Soon, this method turned out impractically and has been displaced by cooling caps which allow a constant cooling of the scalp while easy handling.

However, effectiveness of scalp cooling depends on different factors such as hair texture, chemotherapy regimen, dose of chemotherapy, cooling time, and compliance of the patient.

Recent studies focused on alopecia prevention more than on patients' quality of life and satisfaction. Therefore, data on routine use of cool caps with a focus on efficiency in daily routine and patients' acceptability are missing.

Patient-reported outcomes (PROs) provide results assessed by the use of a patient's report about his or her own health condition "without amendment or interpretation by a clinician or anyone else" and are a valuable source of information when evaluating clinical interventions or treatment toxicity in intervention studies in oncology. PROs can be perfectly used to evaluate the implication of scalp cooling regarding hair preservation but also quality of life outcome which seems even more important.

Women with breast- or gynecological cancer receiving taxane- or anthracycline-based neoadjuvant chemotherapy are included in the study. Chemotherapy can be neoadjuvant, adjuvant or palliative. Up to two lines of chemotherapy are allowed. Scalp cooling with a maintenance temperature of 17°C will be initiated 30 minutes prior to each chemotherapy cycle and stopped 90 minutes after CT. Patients are assessed for alopecia and qualitiy of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast or gynecological cancer planning to undergo CT
* CT can be neoadjuvant, adjuvant or palliative
* Up to two lines of CT are allowed. Adjuvant therapy counts as one line
* CT regime is associated with alopecia
* CT must be planned for at least 4 cycles of taxane or anthracyline-based CT regimen
* written informed consent age 18 and older

Exclusion Criteria:

* Migraine
* Cold allergy/Cold Agglutinins/Morbus Raynaud
* Hematological malignancies (Leukemia, non Hodgkins and other generalized lymphomas)
* Manifest scalp metastases
* Overt cognitive impairment
* Insufficient knowledge of German language

Reference Population:

* Patients with breast or gynecological cancer planning to undergo CT
* CT can be adjuvant, neoadjuvant or palliative
* up to two lines of CT are allowed. Adjuvant therapy counts as one line.
* CT regime is associated with alopecia
* CT must be planned for at least 4 cycles of taxane or anthracycline-based CT regime
* Refuse to undergo scalp cooling
* Patients who have been excluded for the study group for the reason of migraine
* written informed consent
* age 18 and older

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is designed as a clinical trial for women with breast or gyneological cancer, planning to undergo taxane- or anthracyline-based CT in a routine clinical setting.
  For the purpose of comparison, a reference sample is included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Extent of hair preservation | on average of 15 month
  Hair preservation assessed by photo documentation using VAS (Visual Analogue Scale (Grade 1: < 25% hair loss; Grade 2: 25-50% of hair loss; Grade 3: 50-75%)

SECONDARY OUTCOMES:
Assessment of Adverse Events (CTCAE 4.03) | on average of 15 month
  CTCAE are descriptive terminology for reporting adverse events including a grading for each of these adverse events. This 5-point grading has a range from mild symptoms requiring no intervention (grade 1) to life-threatening consequences (grade 4) and finally death (grade 5)
Assessment of patient satisfaction (HAIRDEX) | on average of 15 month
  The Hairdex questionnaire is a reliable and valid instrument for the evaluation of quality of life in patients with hair diseases (i.e. validated in patients with alopecia diffusa and androgenica). Using a five-point Likert Scale (never=0 to always =4), the questionnaire encompasses 48 items composing the 5 subscales symptoms, functioning, emotionals, self-confidence and stigmatization. All scales range from 0-100, higher values indicate higher impairment.
Assessment of quality of life (EORTC) QLQ-C30 | on average of 15 month
  he EORTC QLQ-C30 Aaronson is a self-report measure consisting of 30 items with a 4 point Likert Scale response format. It targets on functioning (physical, role emotional, cognitive, and social functioning and global health/QoL scale) and symptoms (fatigue, nausea and emesis, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhoea, financial difficulties). All scales and single items range from 0-100.
Assessment of quality of life (EORTC) BR23 | on average of 15 month
  The 23-item EORTC QLQ BR23 contains two breast cancer specific functional scales (body image and sexuality) and three symptom scales evaluating arm symptoms, breast symptoms, and systemic therapy symptoms. In addition, we include EORTC single items for hair loss.
Assessment of quality of life (Body Image Scale BIS) | on average of 15 month
  It is a 10 items short instrument suitable for use in clinical trials. The BIS has a single sumscore; the response format is a 4-point Likert scale with high values indicating good body image.
Patient reported-outcomes Common Terminology Criteria for Adverse Events (PRO- CTCAE) | on average of 15 month
  The PRO-CTCAE allow the assessment of those symptoms listed in the CTCAE that can be perceived by a patient him/herself. For most items PRO-CTCAE assesses symptom severity, but for some it covers also symptom frequency and interference with daily activities. In total, this PRO instrument covers 81 symptoms with 126 items using a 5-point Likert scale for grading. For the purpose of this study, we use the PRO-CTCAE-ITEMS (Item Library Version 1.0; Version date: 3/24/2016) Symptom Term: Hair loss.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Marth, Prof Dr, Study Chair — Medical University Innsbruck
Locations (1):
- Medical University Innsbruck, Department of Gynaecology and Obstetrics, Innsbruck, Tyrol, Austria